CLINICAL TRIAL: NCT03838406
Title: A Pilot Trial of Platinum Based Chemotherapy According to BRCA Expressions as First-line Chemotherapy in Patients With Metastatic Gastric Cancer
Brief Title: BReast CAncer Genes(BRCA) Expressions in Metastatic Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung-Ang University (Other)
Responsible Party: Principal Investigator, In Gyu Hwang, Associate Professor, Chung-Ang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1771-001-287
Record Dates: First submitted 2019-02-07; First posted 2019-02-12 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: BRCA Gene Rearrangement
Keywords: Stomach cancer; Chemotherapy; FOLFOX; Capecitabine plus Oxalipatin (CAPOX)
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BRCA1 positive (Experimental): FOLFOX or CAPOX Chemotherapy
  FOLFOX :
  Day 1: Oxaliplatin 85mg/m2 IV + leucovorin 400mg/m2 IV + Fluorouracil (5-FU) 400mg/m2 IV Days 1 and 2: 5-FU 1200mg/m2 IV continuous infusion over 24 hours daily. Repeat cycle every 14 days.
  CAPOX:
  Day 1: Oxaliplatin 130mg/m2 IV Days 1-14: Capecitabine 1000mg/m2 orally twice daily. Repeat cycle every 21 days.
  Interventions: Genetic: BRCA 1; Drug: Chemotherapy
- BRCA1 negative (Active Comparator): FOLFOX or CAPOX Chemotherapy
  FOLFOX :
  Day 1: Oxaliplatin 85mg/m2 IV + leucovorin 400mg/m2 IV + 5-FU 400mg/m2 IV Days 1 and 2: 5-FU 1200mg/m2 IV continuous infusion over 24 hours daily. Repeat cycle every 14 days.
  CAPOX:
  Day 1: Oxaliplatin 130mg/m2 IV Days 1-14: Capecitabine 1000mg/m2 orally twice daily. Repeat cycle every 21 days.
  Interventions: Genetic: BRCA 1; Drug: Chemotherapy

INTERVENTIONS:
Genetic: BRCA 1 — The investigators evaluated the incidence of BRCA loss in patients with advanced gastric cancer and observed the treatment outcome and prognosis.
Drug: Chemotherapy — FOLFOX :
  Day 1: Oxaliplatin 85mg/m2 IV + leucovorin 400mg/m2 IV + Fluorouracil (5-FU) 400mg/m2 IV Days 1 and 2: 5-FU 1200mg/m2 IV continuous infusion over 24 hours daily. Repeat cycle every 14 days.
  CAPOX:
  Day 1: Oxaliplatin 130mg/m2 IV Days 1-14: Capecitabine 1000mg/m2 orally twice daily. Repeat cycle every 21 days.
  Other Names: FOLFOX or CAPOX

SUMMARY:
The investigators evaluated the incidence of BRCA loss in patients with advanced gastric cancer and observed the treatment outcome and prognosis according to BRCA loss. And the investigators evaluated the possibility of BRCA loss as a predictive and prognostic factor.

DETAILED DESCRIPTION:
Stomach cancer is still the leading cause of cancer deaths globally and is reported to be the second leading cause of cancer deaths in Korea (18.7%). Although the number of radical resection has increased due to the development of early diagnosis, many patients experience recurrence after radical resection. It is also diagnosed as a non - resectable disease locally advanced at the time of initial diagnosis, or with a metastasis. In patients with recurrent / metastatic gastric cancer, conventional palliative chemotherapy is the best treatment, and in advanced gastric cancer, combination therapy with fluoropyrimidine (fluorouracil, capecitabine, S1) and platinum (oxaliplatin, cisplatin). The progression-free survival was 3-5 months, and overall survival of 6-10 months in metastatic gastric cancer patients.

The investigators evaluated the incidence of BRCA loss in patients with advanced gastric cancer and observed the treatment outcome and prognosis according to BRCA loss. And the investigators evaluated the possibility of BRCA loss as a predictive and prognostic factor.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic gastric cancer( Adenocarcinoma)
* Eastern Cooperative Oncology Group (ECOG) performance 0-2
* one more measure lesion
* White blood cell count (WBC) > 3000/ul , Platelet > 75,000/ul
* Normal kidney function (serum creatinine < 1.5 ULN)
* Normal Liver function (Aspartate aminotransferase (AST)/ Alanine aminotransferase (ALT) < 3 times of upper normal limit, if liver metastasis, AST/ALT < 5 times of upper normal limit)
* life expectancy is more than 3 months
* Conventional surgery that does not cause the transformation of the target lesion is allowed
* The patient who voluntarily decided to participate in this study and agreed in writing

Exclusion Criteria:

* Her-2 positive advanced gastric cancer
* Central nervous system metastases requiring treatment with symptoms
* Major uncontrolled cardiovascular disease (including myocardial infarction and congestive heart failure within 6 months)
* Uncontrolled infection or other serious diseases
* Patients with serious medical conditions or serious illnesses
* Patient who is pregnant or lactating
* Adjuvant chemotherapy before 6 months (patients who have not received platinum-based chemotherapy even if they are 6 months old can register)
* In the past, if the primary lesion or target lesion was treated with radiation (if the recurred lesion is outside the range of radiation therapy)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate | through study completion, an average of 1 year
  the proportion of patients who have a partial or complete response to therapy; it does not include stable disease and is a direct measure of drug tumoricidal activity.

SECONDARY OUTCOMES:
Progression free survival | through study completion, an average of 1 year
  the time from diagnosis to death by any cause and progression.
Overall survival | through study completion, an average of 1 year
  the time from diagnosis to death by any cause

CONTACTS AND LOCATIONS:
Overall Officials: In Gyu Hwang, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- Chung-Ang University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No